CLINICAL TRIAL: NCT03648450
Title: Feasibility and Acceptability of the Propeller Monitoring System in Children With Persistent Asthma
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Jessica Hollenbach, Assistant Professor of Pediatrics, Connecticut Children's Medical Center
Other Study IDs: Propeller Asthma Study
Record Dates: First submitted 2018-08-09; First posted 2018-08-27 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Propeller Smart Inhaler EMD: All enrolled participants will be given the Propeller Smart Inhaler electronic monitoring device to use for three months to track how often they are using their inhalers either for their regular medication or as a rescue dose.
  Interventions: Other: Propeller EMD

INTERVENTIONS:
Other: Propeller EMD — Propeller electronic monitoring device is a sensor that fits on top of inhalers and uses Bluetooth connection to cell phones to remind patients to take their medication.

SUMMARY:
The main hypothesis of this study is to see if children and adolescents with poorly controlled asthma will find the Propeller electronic monitoring device is feasible and acceptable, and will result in improved medication adherence and asthma control. Preliminary studies indicate that Propeller can improve medication adherence rates in children with asthma and reduce the number of days of reliever medication used. It also has been shown to reduce missed days of school and hospitalizations due to asthma exacerbations. The Propeller device is a sensor that fits over inhalers and uses Bluetooth connection to cell phones to remind patients to take their medication. It also records use of the controller and rescue inhalers, allowing for parents, physicians, and patients to get a fuller and more accurate picture of their adherence to treatment and severity of disease. With improved adherence, asthma control should improve, resulting in a decreased costs and use of services.

DETAILED DESCRIPTION:
This study is a prospective cohort study using a pre-/post-design.

The target population consists of children and adolescents 10-18 years old making an ED visit or admitted to the hospital at Connecticut Children's Medical Center for an asthma exacerbation.

All patients will receive two Propeller devices (for controller and rescue inhalers), an App for their smartphone, and a free Propeller subscription, which provides access support and services, and hardware and software updates. Only the children and adolescents involved with the study will have the app on their phone. The parents will not put the Propeller app on their phone. Families will be asked to share the study information with their primary care provider and will be provided with an introductory letter to bring to the provider, if they so choose.

Data collection will begin at enrollment and will continue through the three-month follow-up period. Propeller provides the option of continuous monitoring and data collection beyond study cessation.

Data uploads to the portal occur automatically for patients and caregivers who have installed the Propeller App on their smartphone. Additionally, patients' primary-care providers will receive a password allowing them to track and access participants' dashboard. Patients will bring a letter to their primary-care provider explaining that they are part of a study of Propeller's device, and receive instructions on how to view the dashboard and adherence data.

At enrollment, participants and parents will complete the Test of Adherence to Inhalers (TAI), Asthma Control Test (ACT) and PedsQL, along with providing baseline medical history/asthma history data and sociodemographic. The TAI, ACT and PedsQL surveys will again be completed one and three months post enrollment information. Additionally, participants will answer an adapted AMDAT survey that will be used to provide acceptability data about the Propeller device.

ELIGIBILITY:
Inclusion Criteria:

1. Children in the ED or inpatient setting presenting with an asthma exacerbation between 10-18 years old
2. History of persistent asthma (defined as prescribed a controller medication)
3. Both the child and primary caregiver/parent have access to a cell phone with an activated number
4. Ability of child's parent/legal guardian to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Child or parent has no access to a personal cell phone.
2. The child has another chronic pulmonary condition (for example, cystic fibrosis)
3. Having any chronic condition that could affect the child's ability to participate in the study (examples: cancer, autism, or cerebral palsy)
4. The subject has an inhaler medication besides the following, given these are the current medications compatible with the Propeller EMD.

   i. Advair HFA ii. Flovent HFA iii. QVAR HFA v. Ventolin HFA vi. ProAir HFA

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The target population consists of children and adolescents 10-18 years old making an ED visit or admitted to the hospital at Connecticut Children's Medical Center for an asthma exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Regular device use at three months | The information will be collected at three months
  This will be assessed by recording the number and percentage of the children and adolescents still using Propeller at three months.

SECONDARY OUTCOMES:
Acceptability of the Propeller EMD as determined by the electronic Medical Devices Assessment Toolkit (AMDAT) | Data will be captured at enrollment, one month and three months after enrollment
  Acceptability will be determined by phone interview and survey response to the modified Adolescent Medical Devices Assessment Toolkit (AMDAT)
Asthma Control | ACT will be assessed at enrollment, one month and three months.
  Asthma control will be measured by the Asthma Control Test (range 0-25 with a higher score representing better asthma control). Change in ACT score will be assessed between baseline and one month and between baseline and three months. A change of 3 or more is considered a clinically significant change.
Device use at one month | The information will be collected at one month
  This will be assessed by recording the number and percentage of the children and adolescents still using the Propeller EMD at one month.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Flores, MD, Study Director — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No